CLINICAL TRIAL: NCT02723552
Title: Trial of Exercise to Prevent HypeRtension in Young Adults
Acronym: TEPHRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Wellcome Trust (Other); Oxford Brookes University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TEPHRA Version 1 16/SC/0016
Record Dates: First submitted 2016-03-16; First posted 2016-03-30 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2016-03

CONDITIONS: Hypertension; Premature Birth
Keywords: preeclampsia; young adult hypertension; preterm birth
MeSH Terms: conditions — Hypertension; Premature Birth; Pre-Eclampsia | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Control participants undergo no intervention.
- Exercise (Experimental): Exercise group participants will undergo 16 weeks of 3x/week supervised aerobic exercise of at least 40 minutes per session. After the supervised exercise phase, they will be monitored and supported to maintain an increased physical activity level for eight months.
  Interventions: Behavioral: Aerobic Exercise

INTERVENTIONS:
Behavioral: Aerobic Exercise — 40 minute aerobic exercise sessions 3x/week.
  Arms: Exercise

SUMMARY:
TEPHRA investigates the effect of exercise on blood pressure and other cardiovascular factors in young adults with different birth histories. TEPHRA will recruit 200 participants from 18-35 years old with elevated blood pressure (100 participants pre-term born and 100 full-term born). Half of the participants from each birth group will be randomised into a 16 week supervised aerobic exercise intervention trial and the other half will be controls.

Participants will complete 3 main study visits:

* Visit 1: Baseline visit conducted at beginning of study
* Visit 2: 16 weeks into study (upon completion of structured exercise intervention for the exercise group)
* Visit 3: End of study (52 weeks) Each visit will repeat the same set of cardiovascular measures including CPET, echo, blood pressure, vascular stiffness, and other measures.

  50 participants from each group will complete an MRI sub-study of the heart, brain, and liver.

DETAILED DESCRIPTION:
DESIGN TEPHRA is a randomized control trial investigating the cardiovascular effects (blood pressure, structure, and function) of aerobic exercise intervention in young adults with elevated blood pressure. The trial will compare outcomes in premature born participants vs full-term born participants.

SCIENTIFIC JUSTIFICATION 1 in 4 adults develop high blood pressure, a risk factor for heart disease and stroke. Although high blood pressure is becoming more common in younger adults, recent literature review shows that most research on exercise and blood pressure has focused on older populations. The effect of exercise on the blood pressure of preterm born young adults has not been well studied or reported. Most babies are born full term (between 37-42 weeks gestation) but 1 in 10 babies are born early (preterm). Evidence suggests that preterm birth may be associated with higher blood pressures and differences in the size, shape and function of the heart and blood vessels. These differences may alter how a person's blood pressure and cardiovascular system respond to exercise. These factors contributed to the investigators pursuing this research study.

The trial is a vehicle to learn more about hypertension in young adults and how exercise helps reduce blood pressure. It will investigate the structure and function of the cardiovascular system and how it responds to exercise. It will specifically seek to improve understanding of how birth histories, such as being born premature may influence blood pressure and response to exercise training.

This trial seeks to illuminate clinically relevant information for one of the most prevalent diseases in the UK (hypertension).

BACKGROUND AND AIMS

1 in 10 babies are born preterm and studies have identified preterm birth to be associated with increased risk of high blood pressure and reduced exercise capacity. This trial aims to advance the understanding of how aerobic exercise affects blood pressure and cardiovascular structure and function in adults aged 18-35 with different birth backgrounds.

PARTICIPANTS:

200 participants (100 preterm born & 100 full term born) aged 18-35 with elevated blood pressure.

RECRUITMENT:

1. Open advertising
2. Hypertension Services at the John Radcliffe Hospital
3. Previous study participants
4. Local GP surgeries

RATIONALE AND FUNDING The study rationale and design has been peer-reviewed to secure external funding from the Wellcome Trust and has been substantially informed by significant interaction with the public and patient involvement group.

ACRONYMS AE Adverse Event CI Chief Investigator CRF Case Report Form CTRG Clinical Trials & Research Governance, University of Oxford GCP Good Clinical Practice GP General Practitioner ICF Informed Consent Form NHS National Health Service PI Principal Investigator PIL Participant/Patient Information Leaflet R&D NHS Trust R&D Department RCT Randomised Control Trial REC Research Ethics Committee SOP Standard Operating Procedure

RECRUITMENT

Participants will be recruited via four approaches:

1. Outpatient Hypertension Clinic, John Radcliffe Hospital, Oxford.
2. Open advertising targeting Oxford residents and students
3. Contacting those who gave consent to be contacted for research from previous ethically approved studies
4. Local GP surgeries

Each approach has been considered from the perspective of the participant and discussed with our public and patient involvement group. Collaboration from the clinical team running the hypertension service will mirror the process used in the YACHT2 study (NHS REC Form Reference:

14/SC/0275 IRAS Version 3.5 Date: 06/05/2014

i)Participant Consent The informed consent process is intended to facilitate participants' understanding of the study. Full study information will be provided to participants in advance of seeking consent, allowing time to interpret the information and ask related questions. Trained study investigators will facilitate the informed consent process. Participants lacking capacity to provide informed consent will be excluded.

ii)Participant Safety Prior to enrollment in the study participants will be given opportunity to fully consider the study procedures. The study team places emphasis on participants understanding that study procedures involve performing a maximal exercise tests and wearing monitoring devices (blood pressure, and physical activity) in their home environments as part of the study. The team will also emphasize that participants will be randomly placed into either the exercise or control group and the exercise group in particular will require a substantial commitment of time and physical effort to complete the 16 week intervention goals. The intervention support team will provide individual guidance and support to the exercise group to support participants in achieving their exercise goals in the safest manner possible. The exercise intervention component is designed at an intensity level (60-80% of max heart rate) and frequency (3 times per week) that is consistent with standard guidelines for safely building aerobic fitness.

Investigators will emphasize that the MRI sub-study involves undergoing magnetic resonance imaging with strong magnetic fields and requires additional screening for contraindications. All participants will be fully screened to ensure there are no contraindications to safely participating in the study. The study procedures are safe and commonly used in both research and clinical practice. Participation in the study does not pose significant risk or burden to the participants.

CONFIDENTIALITY All information and documents collected will be stored securely and kept in strict confidence in compliance with Caldicott Principles and the Data Protection Act.

v)Study samples, investigation results and incidental findings. The use of the participants' study samples and investigations are clearly defined in the participant information leaflet and will be explained during the informed consent process. The investigations used in the study are purely for research purposes but standard operating procedures are in place in the unlikely event of incidental findings that are significant to the participants' well-being. It is possible that some samples will be used for genetic research. The genetic tests would involve looking at common variations in genes that affect how blood vessels work. We do not propose to test for inherited genetic diseases. There is no evidence to suggest that the results of these genetic studies are likely to have significant implications for the participants.

C. Completion of the Study The participant information leaflets and informed consent process clearly explain the intended outcomes of the study and how participant information will be stored. At the end of the study, the study team will coordinate dissemination of data from this study via journal abstracts, articles, and oral/written presentations. Any scientific publications arising from the study will be available on request to all participants as well as a summary of the main findings.

CONSIDERATION OF NULL HYPOTHESES A null hypotheses that "sustained aerobic exercise does not reduce blood pressure in preterm born young adults" was not selected. Rather, studies in older cohorts (birth backgrounds not assessed) strongly suggests that regular aerobic exercise has a blood pressure reducing effect. Previous research has identified differences in the structure and function of the heart and blood vessels of preterm born young adults vs full term born. Accordingly, the hypothesis that "regular aerobic exercise will elicit different blood pressure lowering effects in premature born young adults with elevated blood pressure vs full-term born young adults with elevated blood pressure" will be tested in this study.

SAMPLE SIZE SELECTION Recent systematic review and meta-analysis of randomised control trials identified an average decrease of 5.4mmHg in systolic blood pressure (SBP) post-intervention via supervised exercise in young adults with prehypertension (mean systolic blood pressure at baseline 126 mmHg). The post intervention standard deviation of change was 8.7 mmHg. The investigators' available cross-sectional pilot data suggests that change will be higher in the preterm born participants and participants exposed to maternal hypertension during pregnancy. To calculate the sample size, the investigators used an estimated change of 5 mmHg following 4 months of intervention. The investigators used a SD of 11.3 from the pooled SD for ambulatory systolic blood pressure from cross-sectional pilot data. To observe a treatment effect on systolic blood pressure of 5mmHg, powered to 80% (p=0.05) requires a total sample size of 164 participants. The SD deviation for the pooled 24 hour awake diastolic blood pressure is 8.3 mmHg. To observe a treatment effect on diastolic blood pressure of 5mmHg, powered to 80% (p=0.05) requires a total sample size of 114 participants. The power calculations for systolic blood pressure are used to determine the final sample size, with adjustment to 200 participants to allow for 18% attrition. To ensure primary objectives for the study are answered the study team may recruit additional participants to replace those who drop out of the study.

WHY THE DESIGN AND METHODOLOGY WAS SELECTED The TEPHRA design and methodology was selected to build on two closely related ongoing studies, EXPRESSO and YACHT2 (summarised below). EXPRESSO and YACHT2 collect data that provides significant insight into better characterizing the activity norms and cardiovascular systems of young adults with various birth backgrounds. TEPHRA advances these research themes by employing an intervention arm (aerobic exercise) to investigate the effects of exercise on blood pressure and the structure and function of the cardiovascular system.

JUSTIFICATION FOR INCLUDING A CONTROL ARM Previous studies have identified anatomical and functional differences in the cardiovascular systems of preterm born young adults compared to full-term born controls. The investigators seek to understand the clinical significance of these differences, the response to treatment (in this case exercise) can only be properly assessed by comparing the preterm born cohort against controls.

MINIMISATION OF RESEARCHER EFFECTS AND BIAS

Due to the nature of the intervention (supervised exercise sessions vs "normal" activity levels), TEPHRA is an unblinded trial. However, numerous measures will be taken to minimize investigator effects including:

* All MRI sub-study images will be assessed by investigators who are blinded to participant details

  -- All other images (ie. Ultrasound of heart and small blood vessel imaging) will be assessed by investigators who are blinded to participant details
* Analysis of all blood samples will be completed by laboratories or investigators who are blinded to participant details
* Intervention support protocols are standardised for all participants
* The intervention team field lead (conducts gym visits etc.) is blinded to participant details and does not collect primary study measures

STUDY PROCEDURES AND DATA COLLECTION

SCREENING VISITS Screening Visit Procedures (Visit 0, total time 1 hour) Height, weight, body composition, and blood pressure will be collected. The investigators will also ask candidates to provide information about their medical history and physical activity, and birth history.

* Electrocardiogram (ECG) (20 Minutes) An ECG, will be accomplished to check basic heart function by placing 12 sticky pads on the chest to record the electrical signals the heart makes when it beats. If desired, the investigators will arrange for a candidate's preference of a male or female investigator to set up the ECG. The ECG will take about 20 minutes and will be reviewed by a trained physician. Provided the candidate is happy to continue and there are no exclusionary criteria met, an investigator would then fit the candidate with a 24 hour blood pressure monitor.
* Fitting of 24 hour monitoring equipment (5 minutes) If the screening indicates that the candidate may be a good fit for the trial, the study team will also ask the candidate to wear a blood pressure monitor for 24 hours. It consists of a blood pressure cuff worn on the upper arm that easily fits under clothing. The cuff is attached by a lead to a small box which is slightly larger than a deck of cards. This can be placed in a pocket or attached to a belt provided by the research team. The cuff will inflate and deflates every 30 minutes during the day and every 60 minutes at night to measure blood pressure. It is unlikely that it will disturb sleep and participants are asked to power off the monitor while driving (the research team will show them how to turn the device on and off). A postage paid, addressed envelope will be provided to return the monitor. If all the screening measures indicate that the candidate is a good, safe match for the trail and would like to proceed, the investigators will arrange a convenient time for them to meet for their main trial visits at the Cardiovascular Clinical Research Facility at the John Radcliffe Hospital in Oxford.

MAIN STUDY VISITS COMPLETION OF STUDY VISITS 1-3 (3 hours per visit)

There are three main visits planned for each participant:

* Visit 1: conducted at the beginning of trial (baseline)
* Visit 2: conducted ~16 weeks into trial (this visit coincides with completion of the structured exercise intervention)
* Visit 3: conducted after 52 weeks (at the end of the trial)

Note - If Visit 1 is within 30 days of the screening and the participant has had no change in medical or physical activity status, some basic physical measures (ie. 24 hour blood pressure and body composition) will not be re-assessed. Apart from this noted exception, the same assessments will be repeated at trial visits 1-3. Participants will be asked to have only water for 4 hours before each visit

* Questionnaire (30 minutes) This will collect more detailed information about physical activities and also lifestyle information such as daily routines and use of alcohol and tobacco.
* Physical Measures (15 minutes) (as noted, if the baseline visit is within 30 days of screening, some measures will not be repeated). THe investigators will measure blood pressure and ask participants to walk on the flat for 10 meters while wearing a belt-mounted sensor. The participant will be asked to give a urine sample to test for the presence of protein as an indicator of cardiovascular and blood vessel function related to blood pressure.
* Cardiovascular Measures (45 minutes)

  * Small vessel imaging The investigators will use a special camera to take a picture of the blood vessels in the participants' retina. This is a simple, non-invasive procedure which uses a special camera that looks through the pupil to observe the blood vessels in the back of the eye. This is painless and does not require any physical contact with the eye. The investigators may also use a special microscope to take video images of the small blood vessels on the back of a finger. This is also a painless, non-invasive procedure.
  * Vascular stiffness measurement The investigators will measure stiffness of the blood vessels by placing an inflatable cuff on one arm and also above one knee. This is also a painless, non-invasive procedure.
  * Echocardiogram The investigators will perform an ultrasound (Echocardiogram or "ECHO") of the heart. Participants will be asked to disrobe down to the waist and put on a hospital gown that is untied at the front to allow the study investigators access to place the ultrasound probe on the chest. Participants will lie on a padded treatment table on their left side. The probe is placed on chest and lubricating jelly is used so the probe makes good contact with the skin. Ultrasound waves then create images of the heart on the scanner monitor. The research team are trained to perform echocardiograms, and will ensure that privacy is maintained throughout the visit. Participants can request that a same gender echocardiographer perform the echocardiogram.
* Cardiopulmonary Exercise Testing (50 minutes) During the exercise testing, participants will be asked to donate a total of up to 150mLs (8 to 9 tablespoons) of blood at each trial visit. The blood samples will be stored and analysed for natural compounds and genes involved in blood vessel function and cardiovascular disease development. To allow for collection of blood samples, a cannula will be placed in a vein in the participants' hand or arm. The cannula is a very small, flexible plastic tube that is inserted using a needle and allows for collection of blood without the need for multiple needle pricks. It is also possible to have conventional blood sampling, involving a number of needle pricks, if preferred by the participant.

Exercise testing will allow assessment of heart and lung function during exercise and is the same test used on athletes to see how well they respond to exercise. The exercise test will be performed on a stationary bike. We will ask participants to wear appropriate clothing to exercise in such as shorts or loose fitting track trousers and a comfortable top (hospital scrubs available if needed). Participants will breathe through an opening in a mask worn over their mouth and nose whilst exercising which will allow the measurement of oxygen use and fitness. Participants may stop the test at any time for any reason. As they cycle on the bike, their body response such as heart rate and blood pressure will be recorded. Participants will wear a blood pressure cuff on one arm which will be inflated occasionally throughout the cycle test. The investigators will place three small sticky pads on participants' back to record and ECG during the test.

The exercise testing lasts approximately 10-15 minutes and participants will pedal against gradually increasing resistance. The test is designed to be increasingly difficult as it progresses and will be very physically demanding for the last 3-4 minutes. This is likely to make participants feel quite exhausted, breathe heavily and their leg muscles may ache (particularly if they are not accustomed to exercise). After the test participants will pedal against minimal resistance for a cool down.

--Blood Sampling Before, immediately following, and 20 minutes after the exercise test the cannula in the back of the hand or arm will be used to take a sample of blood. This will allow the study team to measure changes in blood associated with exercising.

DATA MONITORING An independent Data Monitoring Committee will monitor and audit the research project and data collected.

ANALYSIS The analysis will be carried out on the basis of intention-to-treat (ITT). This is, after randomisation, participants will be analysed according to their allocated intervention group irrespective of what they actually receive.

Patient demographic characteristics and other baseline information will be summarised by treatment group. Numbers (with percentages) for binary and categorical variables and mean (standard deviation), or median (interquartile or full range) for continuous variables will be presented. Normality of variables will be assessed by visual assessment of the normality curves and the Shapiro-Wilk test. The analysis of the primary outcome will be assessed using analysis of covariance (ANCOVA) adjusting for baseline values and minimisation factors used in the randomisation process. Results will be presented as adjusted mean difference in change in ambulatory blood pressure between randomised groups at 4 months with 95% confidence intervals (CI) and associated two-sided p value. The analysis of secondary outcomes will also be done using analysis of covariance (ANCOVA) to establish a co-variant model to examine the effect of cardiac structure, vascular function and lifestyle behaviours on exercise capacity. Outcomes measured on more than one occasion will be analysed using a mixed effects model. If the model assumptions are not met and evidence of departure from Normality is observed, transformations of the data will be employed or non-parametric tests will be carried out. Statistical analysis will be carried out using STATA or SPSS statistical software.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, from 18 to 35 years old.
* Verified birth history: preterm birth (<37 weeks) or full-term birth (>37 weeks)
* Ability to access and use computer/internet
* Willing to complete duration of intervention, follow-up and attend study visits at the John Radcliffe Hospital (participants may still withdraw at any time without providing an explanation or rationale)
* 24 hour awake ABP greater than 115/75 mmHg
* Able (in the investigator's opinion) and willing to comply with all study requirements.

Exclusion Criteria:

* Clinic blood pressure greater than 159mmHg systolic and/or 99mmHg diastolic at initial screening
* Pregnancy
* 24 hour awake ABP greater than 150mmHg systolic and/or 95mmHg diastolic
* Clinic blood pressure greater than 140mmHg systolic and/or 90 mmHg diastolic plus evidence of end organ damage secondary to hypertension
* Simultaneous participation in another human or clinical randomized trial (if there is any possibility of compromising health, safety, or well-being, or any possible compromise of study data)
* Unable to walk briskly on the flat for 15 minutes
* Those currently maintaining levels of cardiovascular fitness and activity at or above the levels required for the intervention arm
* Unable to attend the regular supervised exercise sessions
* Use of beta-blockers such as atenolol or equivalent
* BMI >35 kg/m2
* Major contra-indications to exercise participation
* Evidence of cardiomyopathy
* Evidence of inherited cardiac conduction abnormalities
* Evidence of congenital heart disease or significant chronic disease relevant to cardiovascular status

The following are exclusion criteria for the MRI sub-study only:

* a permanent pacemaker • shrapnel injuries
* metal clips in blood vessels of the brain • other metal or electronic implants affected by the magnetic field
* Unsuitable for MRI based on responses on the MRI safety screening form
* an injury to the eye involving fragments of metal

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 203 (Actual)
Dates: Start 2016-06-23 (Actual); Primary Completion 2019-03-29 (Actual); Study Completion 2019-11-26 (Actual)

PRIMARY OUTCOMES:
16 Week Blood Pressure | Measured at baseline and upon completion of 16 week intervention
  Systolic and Diastolic blood pressure measured during 24 hour ambulatory blood pressure at baseline and upon completion of 16 week intervention

SECONDARY OUTCOMES:
52 Week Blood Pressure | Measured at baseline and at 52 weeks post baseline
  Systolic and Diastolic blood pressure measured during 24 hour ambulatory blood pressure at baseline and 52 weeks post randomisation
Peak VO2 | Measured at: - baseline - upon completion of 16 week intervention - 52 weeks post randomisation
  Oxygen uptake and carbon dioxide exchange kinetics across submaximal and peak exercise
Vascular Stiffness | Measured at: - baseline - upon completion of 16 week intervention - 52 weeks post randomisation
  Arterial Pulse Wave Velocity
Cardiac Imaging (3D) | Measured at: baseline - 16 weeks post randomisation - 52 weeks post randomisation
  Cardiac MRI ( MRI subgroup n=100) to assess 3D-shape analysis
Cardiac Imaging (ventricular fxn) | Measured at: baseline - 16 weeks post randomisation - 52 weeks post randomisation
  Cardiac Echocardiography (all participants n=200) 7 Cardiac MRI ( MRI subgroup n=100) to quantify Ventricular Function
Cardiac Imaging (mass) | Measured at: baseline - 16 weeks post randomisation - 52 weeks post randomisation
  Cardiac Echocardiography (all participants n=200) & Cardiac MRI ( MRI subgroup n=100) to quantify cardiac mass
Microvascular Imaging | Measured at: - baseline - upon completion of 16 week intervention - 52 weeks post randomisation
  Dermal and Retinal Capillaroscopy
Blood Analysis | Measured at: - baseline - upon completion of 16 week intervention - 52 weeks post randomisation
  Whole, plasma, and serum blood samples at rest and following peak exercise testing
Brain Imaging (anatomical) | Measured at: baseline - 16 weeks post randomisation - 52 weeks post randomisation
  Brain MRI (MRI subgroup n=100) quantifying ventricular volume and shape
Brain Imaging (lesions) | Measured at: baseline - 16 weeks post randomisation - 52 weeks post randomisation
  Brain MRI (MRI subgroup n=100) quantification of white matter lesions
Brain Imaging (vascular) | Measured at: baseline - 16 weeks post randomisation - 52 weeks post randomisation
  Brain MRI (MRI subgroup n=100) quantification of Vessel Density and Tortuosity
Hepatic Imaging (anatomical) | Measured at: baseline - 16 weeks post randomisation - 52 weeks post randomisation
  Liver MRI (MRI sub-group n=100) anatomocal chara
  * Structure and volume
  * Intra-hepatic lipid content
  * Steatohepatitis
  * Hepatic fibrosis
Hepatic Imaging (fibrosis) | Measured at: baseline - 16 weeks post randomisation - 52 weeks post randomisation
  Liver MRI (MRI sub-group n=100) quantification of hepatic fibrosis
Hepatic Imaging (steatohepatitis) | Measured at: baseline - 16 weeks post randomisation - 52 weeks post randomisation
  Liver MRI (MRI sub-group n=100) quantification of intra-hepatic lipid content
Physical Activity | Measured at: - baseline - upon completion of 16 week intervention - 52 weeks post randomisation
  Objective measure of physical activity (7 day wear of activity monitor) Self-reported questionnaire responses, including self-reported physical activity questionnaires, cognitive and psycho-social questionnaire items and self-efficacy measures.

OTHER OUTCOMES:
Participant Experience | End of Trial
  Optional exit interview of study experience
Economic Evaluation | 36 Month Trial
  Assessment of feasibility for scaling intervention to multi-centre trial including intervention process evaluation by assessing:
  EQ-5D-5L health questionnaire results Structured interviews (study team and personnel) Review of medical notes/GP consultations

CONTACTS AND LOCATIONS:
Overall Officials: Paul M Leeson, Phd, FRCP, Principal Investigator — University of Oxford, Division of Cardiovascular Medicine, Cardiovascular Clinical Research Facility
Locations (1):
- Cardiovascular Clinical Research Facility, Dept of Cardiovascular Medicine, University of Oxford, Oxford, Oxfordshire, United Kingdom

REFERENCES:
- [Background] Bertagnolli M, Luu TM, Lewandowski AJ, Leeson P, Nuyt AM. Preterm Birth and Hypertension: Is There a Link? Curr Hypertens Rep. 2016 Apr;18(4):28. doi: 10.1007/s11906-016-0637-6. PMID 26951245
- [Background] Boardman H, Birse K, Davis EF, Whitworth P, Aggarwal V, Lewandowski AJ, Leeson P. Comprehensive multi-modality assessment of regional and global arterial structure and function in adults born preterm. Hypertens Res. 2016 Jan;39(1):39-45. doi: 10.1038/hr.2015.102. Epub 2015 Sep 24. PMID 26399455
- [Background] Lewandowski AJ, Davis EF, Yu G, Digby JE, Boardman H, Whitworth P, Singhal A, Lucas A, McCormick K, Shore AC, Leeson P. Elevated blood pressure in preterm-born offspring associates with a distinct antiangiogenic state and microvascular abnormalities in adult life. Hypertension. 2015 Mar;65(3):607-14. doi: 10.1161/HYPERTENSIONAHA.114.04662. Epub 2014 Dec 22. PMID 25534704
- [Background] Lewandowski AJ, Bradlow WM, Augustine D, Davis EF, Francis J, Singhal A, Lucas A, Neubauer S, McCormick K, Leeson P. Right ventricular systolic dysfunction in young adults born preterm. Circulation. 2013 Aug 13;128(7):713-20. doi: 10.1161/CIRCULATIONAHA.113.002583. PMID 23940387
- [Derived] Lapidaire W, Forkert ND, Williamson W, Huckstep O, Tan CM, Alsharqi M, Mohamed A, Kitt J, Burchert H, Mouches P, Dawes H, Foster C, Okell TW, Lewandowski AJ, Leeson P. Aerobic exercise increases brain vessel lumen size and blood flow in young adults with elevated blood pressure. Secondary analysis of the TEPHRA randomized clinical trial. Neuroimage Clin. 2023;37:103337. doi: 10.1016/j.nicl.2023.103337. Epub 2023 Jan 24. PMID 36709637
- [Derived] Burchert H, Lapidaire W, Williamson W, McCourt A, Dockerill C, Woodward W, Tan CMJ, Bertagnolli M, Mohamed A, Alsharqi M, Hanssen H, Huckstep OJ, Leeson P, Lewandowski AJ. Aerobic Exercise Training Response in Preterm-Born Young Adults with Elevated Blood Pressure and Stage 1 Hypertension: A Randomized Clinical Trial. Am J Respir Crit Care Med. 2023 May 1;207(9):1227-1236. doi: 10.1164/rccm.202205-0858OC. PMID 36459100
- [Derived] Williamson W, Lewandowski AJ, Huckstep OJ, Lapidaire W, Ooms A, Tan C, Mohamed A, Alsharqi M, Bertagnolli M, Woodward W, Dockerill C, McCourt A, Kenworthy Y, Burchert H, Doherty A, Newton J, Hanssen H, Cruickshank JK, McManus R, Holmes J, Ji C, Love S, Frangou E, Everett C, Hillsdon M, Dawes H, Foster C, Leeson P. Effect of moderate to high intensity aerobic exercise on blood pressure in young adults: The TEPHRA open, two-arm, parallel superiority randomized clinical trial. EClinicalMedicine. 2022 May 13;48:101445. doi: 10.1016/j.eclinm.2022.101445. eCollection 2022 Jun. PMID 35706495
- [Derived] Williamson W, Huckstep OJ, Frangou E, Mohamed A, Tan C, Alsharqi M, Bertagnolli M, Lapidaire W, Newton J, Hanssen H, McManus R, Dawes H, Foster C, Lewandowski AJ, Leeson P. Trial of exercise to prevent HypeRtension in young adults (TEPHRA) a randomized controlled trial: study protocol. BMC Cardiovasc Disord. 2018 Nov 6;18(1):208. doi: 10.1186/s12872-018-0944-8. PMID 30400774